CLINICAL TRIAL: NCT04779099
Title: Pilot Randomized Controlled Trial of a Brief Psychological Intervention for Suicidal Patients with Borderline Personality Disorder in the Emergency Department
Brief Title: Trial of a Brief Psychological Intervention for Suicidal Patients with Borderline Personality Disorder in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Anne Sonley, Psychiatrist and Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-796
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Borderline Personality Disorder; Suicide and Self-harm
MeSH Terms: conditions — Borderline Personality Disorder; Suicide; Self-Injurious Behavior | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4-session intervention (Experimental)
  Interventions: Behavioral: Brief 4-session intervention for borderline personality disorder; Behavioral: Treatment as usual
- Treatment as usual (Active Comparator)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Brief 4-session intervention for borderline personality disorder — Intervention consists of weekly 50-minute 1:1 sessions focused on psycho-education, here-and-now problem solving and safety planning. One of the sessions can involve a significant other to provide psychoeducation about the disorder and to facilitate support. This intervention is detailed in a published manual.
  Arms: 4-session intervention
Behavioral: Treatment as usual — TAU comprises access to psychiatric assessment, medication review, and unscheduled sessions with allied health professionals using a drop-in model of care.

SUMMARY:
When in crisis, people with borderline personality disorder (BPD) frequently seek care in emergency departments (EDs) often presenting with suicide and self-harm behaviour. There is no established evidence-based brief intervention for patients with BPD in ED settings, however a 4-session psychotherapeutic intervention for people with personality disorders in ED settings was tested in Australia and showed promising results in reduced health care utilization. The proposed pilot randomized controlled trial will assess the feasibility of delivering this 4-session intervention in the ED for people with BPD who present with suicidal ideation or self-harm with the aim of reducing health care utilization.

ELIGIBILITY:
Inclusion Criteria:

1. aged 16 or older
2. presenting to ED with self-harm and/or suicidal ideation; and
3. meeting criteria for BPD on the Structured Clinical Interview for DSM-5 Personality Disorders

Exclusion Criteria:

1. unable to give informed consent;
2. meeting DSM-5 criteria for severe substance use disorder, schizophrenia spectrum disorder or bipolar disorder I mania based on the Structured Clinical Interview for DSM-5 (28); and/or
3. IQ < 70 based on the Wechsler Test of Adult Reading

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Primary clinical outcome measure - Emergency Department Visits | 1, 3 and 6 month follow up
  The primary clinical outcome will be the mean group difference in frequency of ER visits on the Client Service Receipt Inventory (CSRI)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided